CLINICAL TRIAL: NCT06916078
Title: A Phase 1, Multicenter, Sequential-Design, Single-Dose, Open-Label Study of Lepodisiran in Participants With Normal Hepatic Function and Participants With Mild, Moderate, or Severe Hepatic Impairment
Brief Title: A Study of Lepodisiran (LY3819469) in Participants With Normal, Mild, Moderate, or Severe Liver Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 27200; J3L-MC-EZEH (Other: Eli Lilly and Company); 2024-520315-40-00 (Other: EU CT)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Liver Dysfunction; Healthy
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lepodisiran Group 1 (Experimental): Lepodisiran administered subcutaneously (SC)
  Interventions: Drug: Lepodisiran
- Lepodisiran Group 2 (Experimental): Lepodisiran administered SC
  Interventions: Drug: Lepodisiran
- Lepodisiran Group 3 (Experimental): Lepodisiran administered SC
  Interventions: Drug: Lepodisiran
- Lepodisiran Group 4 (Experimental): Lepodisiran administered SC
  Interventions: Drug: Lepodisiran

INTERVENTIONS:
Drug: Lepodisiran — Lepodisiran administered SC
  Other Names: LY3819469

SUMMARY:
The main purpose of this study is to evaluate how much lepodisiran gets into the blood stream and how long it takes the body to get rid of it when given as a subcutaneous (SC) injection under the skin to participants with mild, moderate, or severe liver function impairment compared to participants with normal liver function. The study will also evaluate how well lepodisiran is tolerated and what side effects may occur in these participants.

The study will last up to approximately 9 weeks, excluding screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight of 55 kilogram (kg) or more and body mass index within the range 19.0 to 42.0 kilogram per square meter (kg/m²)
* Additional Inclusion Criteria for Participants Without Hepatic Impairment in Group 1:

  * Healthy participants with clinically normal hepatic function
* For Participants with Mild to Severe Hepatic Impairment in Groups 2 through 4:

  * Participants with hepatic impairment classified as Child-Pugh score A, B, or C (mild, moderate, or severe impairment). Diagnosis of chronic hepatic impairment of greater than 6 months, per physician diagnosis and standard-of-care practice

Exclusion Criteria:

* Have significant history of, or current, cardiovascular (CV), respiratory, hepatic (hepatic applies to Group 1 only), renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Have severe atopy or a history of clinically significant multiple or severe drug allergies
* Have known allergies to lepodisiran, related compounds, or any components of the formulation
* Have a history of, or current, psychiatric disorders
* Have had any malignancy within the past 5 years
* Have estimated glomerular filtration rate (eGFR) less than 60 milliliters per minute per 1.73 m² (mL/min/1.73 m²) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Have participated, within the last 1 month, in a clinical study involving an investigational product

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Lepodisiran | Baseline Up to 9 weeks
  PK: AUC of Lepodisiran
PK: Maximum Concentration (Cmax) of Lepodisiran | Baseline Up to 9 weeks
  PK: Cmax of Lepodisiran

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
- CRU Early Phase Unit, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/591635